Phone: (+84) 28 3855 4269 – Fax: (+84) 28 3950 6126 Website: www.bvdaihoc.com.vn – Email: bvdh@umc.edu.vn



Ver5:12062023

## PARTICIPANT INFORMATION SHEET

### 1. Background Information

Research Title: Characterization Of Vietnamese Patients With Obesity At Outpatient Clinics

### **Executor:**

• Topic leader: Tran Quang Nam, MD. PhD.

• Topic co-chair: Hoang Khanh Chi, MD.

## 2. What is the purpose of this study?

- Description of population characteristics and awareness of obese patients at the outpatient clinic of University Medical Center Ho Chi Minh City and My Duc General Hospital.

## 3. Why was I invited to participate in this study?

- You are invited to participate in this study based on the initial assessment of body mass index more than 25 kg/m<sup>2</sup>, equivalent to the standard obesity classification for the Asia-Pacific population.

## 4. What do I need to do to participate in this study?

- You need to follow the steps in the research, including: (1) having your anthropometric measurements taken according to the standard procedure in the study, and (2) answering the questions in the data collection form from the researchers.

# 5. What are my responsibilities when participating in research?

- You need to strictly follow the doctor's instructions and follow all the steps in the treatment and research process as described above.

## 6. What are the possible risks and disadvantages of the study?

- This is a descriptive study, without intervention in patients, so there are no risks and disadvantages for study participants.

215 Hong Bang, Ward 11, District 5, HCMC Phone: (+84) 28 3855 4269 – Fax: (+84) 28 3950 6126

Website: www.bvdaihoc.com.vn - Email: bvdh@umc.edu.vn



Ver5:12062023

- You will not have to pay any additional costs for participating in the study. If you do not agree to participate in the study, you can continue with the treatment as usual without any

problems.

7. What are my rights and benefits for participating in this study?

- You will be measured your height, weight, body mass index (BMI), and body fat mass

(BIA) for free (the cost of this service is 100,000 Vietnam Dong).

- You will be consulted on your obesity status and initial intervention.

- Your participation in the study will contribute to the development of epidemiological data

and characteristics of the obese population in Vietnam, which will be meaningful in the

development of obesity studies in the country and in the Southeast Asia region in the future.

8. Confidentiality

- The information and research data collected from participating in the study will be kept

confidential by the researcher by encryption.

9. Not participating in the study

- Your choice to participate in the study is voluntary.

- If you have been admitted to the study but change your mind, you can withdraw from the

study at any time. You will still be cared for and treated according to the hospital's

regulations.

10. Treatment and research costs

- You will not be paid for your participation in the study. You will pay for your own

medical expenses according to the routine procedure.

11. Who do you contact if you need information?

- If you have any questions regarding the research, please contact: Hoang Khanh Chi,

phone number: (+84)-985578494





Ver5:12062023

### **INFORMED CONSENT**

Research name: Characterization Of Vietnamese Patients With Obesity At Outpatient Clinics

#### **Executor**

- **Topic leader**: Tran Quang Nam, MD. PhD.
- **Topic co-chair:** Hoang Khanh Chi, MD.

### PARTICIPANT'S CONFIRMATION

I read the information provided about the study in the Participant Information Sheet about the study and the Informed Consent Form. I was well-explained by the researchers about the study and the procedures for volunteering to participate in the study. I have had the opportunity to ask questions about the research and I am satisfied with the answers given. I had the time and opportunity to consider participating in this study. I have understood that I have a right to access to the information described in the Participant Information Sheet. I understand that I have the right to withdraw from the study at any time for any reason. I agree that the doctors who are treating me (if any) will be notified of my participation in the study.

| for any reason. I agree that the doctors warticipation in the study. | who are treating me (if any) | will be notified of my |
|---|---|---|
| Participant's name | Signature | Day |
| I, the undersigned, hereby declare study participants. Participants clearly benefits of participating in blood tests an | that I have fully explained understood the purposes, p | the information to the |
| Researcher's name | Signature | Day |